CLINICAL TRIAL: NCT05219149
Title: Exploring Factors in Patient and Family Consideration of Treatment for Pediatric Central Nervous System Tumors
Brief Title: CNS Qualitative Interview
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Other Study IDs: 21-3870.cc; NCI-2021-14424 (Other: CTRP)
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Central Nervous System Cancer
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with CNS Tumors: feasibility study of family interviews of those who are making decisions about treatment for newly diagnosed or relapsed CNS tumors. For patients 12 years of age and younger, caregivers only will be included in the interviews. For patients 13-17 years of age, caregivers will have the option to include the patient in the interviews. For patients 18 years of age and older, patients will have the option to include their caregivers in the interviews.
  Interventions: Behavioral: Qualitative Interviews

INTERVENTIONS:
Behavioral: Qualitative Interviews — Conduct qualitative interviews with patients and families who are considering treatment options for new or recurrent CNS tumors to identify specific barriers to full participation in treatment and clinical trial enrollment (e.g., transportation, childcare, ancillary expenses). Qualitative interviews will be structured to comprehensively address potential barriers but also open-ended to give patients and families freedom to discuss a wide range of challenges.

SUMMARY:
Explore factors involved in decision making for patients with new or recurrent CNS tumors and their families surrounding treatment planning and clinical trial enrollment.

DETAILED DESCRIPTION:
Explore factors involved in decision making for patients with new or recurrent CNS tumors and their families surrounding treatment planning and clinical trial enrollment. The team will conduct qualitative interviews with a diverse group of patients and families considering treatment for new and recurrent CNS tumors to determine challenges surrounding treatment and study enrollment that may be modifiable through community, hospital, and University of Colorado Cancer Center resources. The team will then assess the impact of these resources on decision making through follow-up interviews.

ELIGIBILITY:
Inclusion Criteria:

1. Be the parent or caregiver of a child or young adult receiving treatment at CHCO

   a. Child must meet one criterion below: i. Newly diagnosed with a CNS tumor ii. Relapse of a CNS tumor requiring further therapy. Therapy may be standard of care of dictated by an open clinical trial
2. Patient 18 years of age or older a. Must meet one of the criteria below: i. Newly diagnosed with a CNS tumor ii. Relapse of a CNS tumor requiring further therapy. Therapy may be standard of care of dictated by an open clinical trial

Exclusion Criteria:

* Does not meet inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parents and caregivers will be eligible for participation if their child is newly diagnosed with or has had a recent relapse of a CNS tumor that will require further therapy. Therapy may be either standard of care or dictated by an open clinical trial.
  For patients 12 years of age and younger, caregivers only will be included in the interviews. For patients 13-17 years of age, caregivers will have the option to include the patient in the interviews. For patients 18 years of age and older, patients will have the option to include their caregivers in the interviews.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-23 (Estimated)

PRIMARY OUTCOMES:
Identify barriers to trial enrollment | 12 months
  Qualitative interviews with patients and families who are considering treatment options for new or recurrent CNS tumors to identify specific barriers to full participation in treatment and clinical trial enrollment (e.g., transportation, childcare, ancillary expenses). Qualitative interviews will be structured to comprehensively address potential barriers but also open-ended to give patients and families freedom to discuss a wide range of challenges.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Green, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided